CLINICAL TRIAL: NCT04438486
Title: Effects of Barley Green in Patients With Hyperuricemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Jinhua Municipal Central Hospital (Other); Quzhou Kecheng People's Hospital (Unknown); First Affiliated Hospital of Wenzhou Medical University (Other); Zhejiang Cancer Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-411
Record Dates: First submitted 2020-06-17; First posted 2020-06-18 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-07

CONDITIONS: Dietary Supplement

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dietary advice (Active Comparator)
  Interventions: Behavioral: Group A
- dietary advice+ Barely Green (Experimental)
  Interventions: Dietary Supplement: Group B

INTERVENTIONS:
Behavioral: Group A — specific dietary advice for Hyperuricemia
  Arms: dietary advice
Dietary Supplement: Group B — Barely Green（three times a day, 5g(10 tablets)） dietary advice for Hyperuricemia as Group A
  Arms: dietary advice+ Barely Green

SUMMARY:
This experiment evaluates the effect of Barley Green in patients with hyperuricemia ， and explores the effect of Barley Green on metabolic indexes such as uric acid, blood lipids, blood glucose, free fatty acids。130 adult participants , age 18 to 65 years, will be randomized into one of the two arms. Arm A (control group) will receive dietary guidance. Arm B will receive dietary guidance and Barley Green.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old those who are willing to accept assessment and sign informed consent.
* Under the normal purine diet, two fasting blood uric acid levels on different days: 420umol/l <blood uric acid <540 umol/l (male), 360 umol/l <blood uric acid <540 umol/l (female)

Exclusion Criteria:

* Patients currently receiving treatment for hyperuricemia；
* Suffering from diseases that affect the digestion and absorption(such as chronic diarrhea, constipation, severe gastrointestinal inflammation, active gastrointestinal ulcers, after gastrointestinal resection, cholecystitis/cholecystectomy, etc.)；
* Suffering from cardiovascular and cerebrovascular diseases, grade 3 hypertension, chronic hepatitis, malignant tumors, anemia, mental illness and memory disorders, epilepsy and other diseases;
* At the same time receive other functional food nutrition support (plant active substances, health food);
* Patients with abnormal liver function (alanine aminotransferase or/and aspartate aminotransferase exceeds 3 times the upper limit of normal value); patients with abnormal renal function (serum creatinine exceeds the upper limit of normal value)；
* Suffering from infectious diseases such as active tuberculosis and AIDS;
* People who are severely allergic to the ingredients of research；
* During pregnancy or lactation;
* Patients with physical disabilities and clinicians think it is not suitable to participate in the study (for example, suffering from serious diseases not included in the discharge criteria)；
* Gouty arthritis attack ≥ 2 times;
* One episode of gouty arthritis with blood uric acid >480 umol/l, or any of the following: age <40 years old, evidence of gout stone or urate deposition in the joint cavity, uric acid nephrolithiasis or renal impairment (GFR≤89ml/(min·1.73m2)), hypertension, impaired glucose tolerance or diabetes, dyslipidemia, obesity, coronary heart disease, stroke, cardiac insufficiency;
* Blood uric acid>480 umol/l combined with any of the following: uric acid nephrolithiasis or renal impairment (GFR≤89ml/(min·1.73m2)), hypertension, impaired glucose tolerance or diabetes, dyslipidemia, obesity, Coronary heart disease, stroke, heart failure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
uric acid level | 3 months

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang cancer hospital, Hangzhou, Zhejiang
  - Jinhua municipal central hospital, Jinhua, Zhejiang
  - Quzhou Kecheng People's Hospital, Quzhou, Zhejiang
  - The first affiliated hospital of Wenzhou medical university, Wenzhou, Zhejiang
  - Beijing Shijitan Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided